CLINICAL TRIAL: NCT06441747
Title: Phase II Study of the Combination of Durvalumab (MEDI4736) (PDL1 Inhibitor) and Olaparib (PARP Inhibitor) in Advanced Cholangiocarcinoma After Initial Chemotherapy and Durvalumab (BIL-PPP)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Collaborators: Wayne Elphinstone Research Fund (Unknown); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIL-PPP
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cholangiocarcinoma
Keywords: Advanced Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — durvalumab; olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab and Olaparib (Experimental): This is a trial of Durvalumab in combination with olaparib. Durvalumab will be administered at a dose of 1500mg intravenously every 4 weeks. Olaparib will be administered orally at a dose of 300mg twice daily continuously. This combination will be administered for a maximum of two years unless unacceptable toxicities or progressive disease.
  Interventions: Drug: Durvalumab; Drug: Olaparib

INTERVENTIONS:
Drug: Durvalumab — Durvalumab will be administered at a dose of 1500mg intravenously every 4 weeks.
  Other Names: Imfinzi
Drug: Olaparib — Olaparib is administered at a dose of 300mg bd in a continuous 28-day cycle. On day 1 of each cycle, the morning dose of Olaparib should be taken no more than 1 hour prior to infusion of durvalumab. It is expected that patients will receive up to 24 months of a combination of olaparib and durvalumab, or until disease progression, unacceptable toxicities, or withdrawal of consent.
  Other Names: Lynparza

SUMMARY:
The aim of this study is to investigate whether the combination of durvalumab and olaparib in the maintenance setting after initial chemotherapy and durvalumab will benefit patients with locally advanced or metastatic cholangiocarcinoma.

DETAILED DESCRIPTION:
The primary objectives are

(i) To describe the efficacy of PARPi and PDL1 inhibition in the maintenance setting of metastatic cholangiocarcinomas.

(ii) To refine selection of the patient population who are most likely to benefit from the combination of PDL1 (Durvalumab) and PARP (Olaparib) inhibition in the maintenance setting following initial chemotherapy (cisplatin + gemcitabine + Durvalumab) (post hoc translational analysis).

The secondary objectives are (i) To evaluate toxicity of the combination of durvalumab and olaparib. (ii) To evaluate progression-free and overall survival with the combination of durvalumab and olaparib (PFS, OS).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, and life expectancy>12 weeks
2. Weight: >30kg
3. Histologically proven locally advanced or metastatic/unresectable cholangiocarcinoma
4. Documentation of RECISTv1.1 measurable disease
5. Must not have had radiologic progression after 6-8 cycles of gemcitabine and cisplatin and durvalumab
6. Adequate haematological and end-organ function as defined by the following parameters:

   1. Haemoglobin ≥ 90g/L (without a transfusion in the past two weeks)
   2. Platelets ≥100 x 109/L (without a transfusion in the past two weeks)
   3. Neutrophils ≥ 1.0 x 109/L (without the use of G-CSF in the 4 weeks prior to first dose)
   4. ALT/AST <3x ULN irrespective of presence of liver metastases
   5. Serum bilirubin ≤ 1.5x ULN except in cases of known Gilbert's Syndrome where total bilirubin must be <4x ULN
   6. Albumin ≥ 25 g/L
   7. Serum Creatinine ≤1.5 x ULN or eGFR ≥ 30mL/min/1.73m2 as calculated by Cockcroft Gault Equation
7. Able to swallow oral medications without any difficulties or medical history associated with malabsorption or any conditions that may impact on compliance or absorption of the study treatment.
8. Women of Childbearing potential must be either totally abstinent or agree to use at least one highly effective method of birth control (e.g., oral contraceptive pill, barrier method) for the duration of the study and for at least 6 months after the final dose of study medication. They must also have a negative serum beta-hCG in the 7 days prior to first dose of study drug.
9. Non-sterile males and their female partners must also either be totally abstinent or agree to use at least one highly effective method of birth control (e.g., oral contraceptive pill, barrier method) for the duration of the study and for at least 6 months after the final dose of study medication.
10. Patient is willing and able to comply with the protocol for the duration of the study, including undergoing treatment and scheduled visits and examinations including follow up.
11. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

1. Previous use of a PARP inhibitor.
2. All prior treatment-related AEs must have resolved to a CTCAE v5 Grade 1 or less prior to commencement of study medication, with the exception of alopecia and peripheral neuropathy which can be grade 2 or less.

   i. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.

   ii. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or olaparib may be included only after consultation with the Study Chairs.
3. Known symptomatic or progressive CNS metastases or leptomeningeal disease. Patients with treated brain metastases are eligible for inclusion in the study if they had received treatment >4 weeks prior to commencement of study medication, and have a repeat MRI scan demonstrating stability in disease.
4. Patients with severe chronic or active infections requiring systemic antibiotics or antifungals in the two weeks prior to starting trial treatment.
5. Any of the following cardiovascular risk factors:

   1. Acute myocardial infarction (MI) ≤6 months prior to study registration
   2. New York Heart Association (NYHA) Heart Failure Class III-IV within ≤6 months of registration
   3. History of cerebral vascular accident (CVA) within 6 months of first dose
6. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study, or during the follow-up period of an interventional study.
7. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
8. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
9. History of allogeneic organ transplantation.
10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia.
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
    3. Any chronic skin condition that does not require systemic therapy.
    4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
    5. Patients with celiac disease controlled by diet alone.
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhoea, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs, or compromise the ability of the patient to give written informed consent.
12. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of IP and of low potential risk for recurrence.
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
    3. Adequately treated carcinoma in situ without evidence of disease.
13. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
14. History of active primary immunodeficiency.
15. Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of anti HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

    1. Participants co-infected with HBV and HCV, or co-infected with HBV and HDV, namely: HBV positive (presence of HBsAg and/or anti HBcAb with detectable HBV DNA); AND
    2. HCV positive (presence of anti-HCV antibodies); OR
    3. HDV positive (presence of anti-HDV antibodies).
16. Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice). Known HIV infection that is not well controlled. All of the following criteria are required to define an HIV infection that is well controlled: undetectable viral RNA load for 6 months prior, CD4+ count of >500, no history of AIDS-defining opportunistic infection within the past 12 months, and stable for at least 6 months on the same anti-HIV medications.
17. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection)
    2. Systemic corticosteroids at physiologic doses that do not exceed 10 mg/day of prednisolone or its equivalent.
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
18. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 90days after the last dose of IP.19. Female patients who are pregnant or breastfeeding, or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.

20. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

21. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 12 months post randomisation
  To describe the efficacy of PARPi and PDL1 inhibition in the maintenance setting of metastatic cholangiocarcinomas.
Evaluate benefit | 12 months post randomisation
  To refine selection of the patient population who are most likely to benefit from the combination of PDL1 (durvalumab) and PARP (olaparib) inhibition in the maintenance setting following initial chemotherapy (cisplatin + gemcitabine + durvalumab) (post hoc translational analysis).

SECONDARY OUTCOMES:
Evaluate toxicity | 12 months post randomisation
  To evaluate toxicity of the combination of durvalumab and olaparib.
Progression free survival | 12 months post randomisation
  To evaluate progression-free survival with the combination of durvalumab and olaparib (PFS).
Overall survival | 12 months post randomisation
  To evaluate overall survival with the combination of durvalumab and olaparib (OS).

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (8):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Monash Medical Centre, Clayton, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Austin Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No